CLINICAL TRIAL: NCT04227496
Title: Evaluating the Effect of Auditory Disturbances on Human Movement
Brief Title: The Effect of Auditory Disturbances on Human Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FOU-UU-2018-194_Sub-project1
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Noise1 (Active Comparator): A sound will be played while moving a body part through range of motion
  Interventions: Device: Auditory disturbances
- Noise2 (Active Comparator): A sound (different from Noise 1) will be played while moving a body part through range of motion
  Interventions: Device: Auditory disturbances
- No noise (No Intervention): No sound will be played while moving a body part through range of motion

INTERVENTIONS:
Device: Auditory disturbances — A sound will be played from a portable device (smartphone) during movement
  Arms: Noise1; Noise2

SUMMARY:
This study sets out to investigate the potential effect of auditory disturbances on human movement

DETAILED DESCRIPTION:
Clinicians routinely investigate/test human movement but if/how this is effect by auditory disturbances is unclear. This study sets out to investigate the impact of auditory disturbances on human movement.

ELIGIBILITY:
Criteria:

Inclusion Criteria: - Healthy participants

* Pain free healthy participants
* Able to speak, read and understand Danish and English

Exclusion Criteria: - Healthy participants

* Pain from the neck, back, arm or leg during the past 6 months up to the test session
* Former surgery in neck, back, arm or leg restricting normal movement
* Current or previous chronic or recurrent pain condition
* Pregnancy
* Current or previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate

Inclusion Criteria: - Pain population

* Self reported ongoing or recurring pain from neck, back, arm or leg
* Able to speak, read and understand Danish and English

Exclusion Criteria: - Neck pain population

* Current or previous chronic or recurrent pain condition
* Former surgery in neck, back, arm or leg restricting normal movement
* Pregnancy
* Current or previous neurologic, musculoskeletal (other than what is included) or mental illnesses
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-13 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion | During a single test session (approximately 2hours)
  Range of movement will be assessed by measuring displacement of the body part being moved (i.e. moving the head, back, arm or leg from a neutral position to end of range in flexion, extension, rotation, addiction or abduction)

SECONDARY OUTCOMES:
Experienced pain | During a single test session (approximately 2hours)
  Any potential pain during the functional tasks will be monitored using a 0-11 numeric rating scale (NRS) with 0 being no pain and 10 being worst imaginable pain
Experienced difficultness of performing movement | During a single test session (approximately 2hours)
  a 6-point Likert scale going from 0 = 'no problems',
  1 = minimally difficult; 2 = somewhat difficult; 3 = fairly difficult; 4 = very difficult; 5 = unable to perform

CONTACTS AND LOCATIONS:
Overall Officials: Steffan WM Christensen, PhD, Principal Investigator — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- Department of Physiotherapy, University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No